CLINICAL TRIAL: NCT03665025
Title: Immediate Implant Placement With Immediate Professionalization in the Maxillary Esthetic Zone Using Mixture of Allograft and Xenograft vs Xenografts to Augment the Jumping Gap
Brief Title: Immediate Implant Placement With Immediate Professionalization in Aesthetic Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohammed nashmi hammad, Lecturer of oral and maxillofacial surgery-Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14422017463550
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Implant Site Reaction
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: jumping gap area in aesthetic area
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant placement with xenograft (Experimental): Immediate implant placement with the use of xenograft as grafting material
  Interventions: Other: immediate implant using mixed allograft and xenograft
- immediate implant using mixed allograft and xenograft (Experimental): Immediate implant placement with using mixture of allograft and xenograft material
  Interventions: Other: immediate implant using mixed allograft and xenograft

INTERVENTIONS:
Other: immediate implant using mixed allograft and xenograft — immediate implant using mixed allograft and xenograft in anterior area to fill jumping area

SUMMARY:
Immediate implant placement with immediate professionalization in the maxillary esthetic zone using mixture of allograft and xenograft vs xenografts to augment the jumping gap

DETAILED DESCRIPTION:
Implant placement in fresh extraction sockets in conjunction with appropriate guided bone regeneration has many benefits, which ultimately affect the total treatment plan. The immediate placement of implants provides significant advantages, including fewer surgical procedures, shorter treatment time, and improved esthetics. The goals of osseous replacement are maintenance of contour, elimination of dead space, and reduce postoperative infection, provide good support for dental implant and enhance bony and soft tissue healing. allograft bone has gold standard over other augment techniques including favorable bone quality and minimal bone resorption.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with badly broken teeth in upper esthetic zone indicated for extraction, presence of at least 4 mm of bone beyond the root apex to guarantee implant primary stability, implant placement within the alveoli confines.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Presence of fenestrations or dehiscence of the residual bony Walls after extraction.
* Heavy smokers more than 20 cigarettes per day .(24)
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Crestal bone loss | 1 year
  Will be measured using calliper with scale(1-10mm) for evaluation of crestal bone loss around implant which are the lower values represent a better outcome.

SECONDARY OUTCOMES:
Patient satisfaction | 1 year
  Will be measured using a satisfaction table chart which divided in 4 paraments with scale from 1-4 include( pain-infection-radiography-successful implant ),the number represent (4 excellent-3 very good -2 good-1 bad)

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed, Kuwait City, Q8, Kuwait